CLINICAL TRIAL: NCT03682016
Title: The Effect of Central Blood Pressure on Clinical Outcome in Diabetic Hypertensive Patients in Assiut University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Nader Ramzy Tamer, principle investigator, Assiut University
Other Study IDs: Assiut 93
Record Dates: First submitted 2018-07-26; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Central Blood Pressure in Diabetic Hypertensive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent decades, some observational studies suggest that peripheral BP measured by brachial artery may not necessarily represent BP measured in the aortic artery which is known as central BP .In addition, some clinical trials also revealed that despite with comparable peripheral BP, patients with high central BP had significantly higher cardiovascular risk compared with those with low central BP indicating that central BP might be an independent predictor for CVD

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is amajor risk factor for cardiovascular and renal diseases[1] .It is known about two thirds of diabetic patients died from these complication .Numerous epidemiological studies demonstrate that DM is commonly accompanied with hypertension and patients with diabetes and hypertension have higher renal and cardiovascular risks compared with those with either hypertension or diabetes. Therefore, better evaluating and managing BP in diabetic patients with hypertension is clinically relevant.

Hypertension also is a major risk factor for cardiovascular diseases (CVD) and all-cause mortality . Numerous randomized controlled trials using antihypertensive drugs and meta-analysis demonstrate that lowering peripheral blood pressure (BP) is beneficial for reducing cardiovascular and renal events.

In recent decades, some observational studies suggest that peripheral BP measured by brachial artery may not necessarily represent BP measured in the aortic artery which is known as central BP.

In addition, some clinical trials also revealed that despite with comparable peripheral BP, patients with high central BP had significantly higher cardiovascular risk compared with those with low central BP indicating that central BP might be an independent predictor for CVD

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 - 60 years old
* Patients in group A and B are documented to have type 2 DM
* Patients in group A are documented to have essential hypertension .
* Hypertensive patients enrolled must be compliant on their treatment for at least one month

Exclusion Criteria:

* Pregnancy or breastfeeding .
* Concomitant therapy of digoxin, lithium, non-depolarizing skeletal muscle relaxants, sex hormone .
* Documented rheumatic diseases such as systemic lupus erythematosus .

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 150 patients attending internal medicine clinics in Assiut University Hospitals
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
relation between central systolic blood pressure and the risk of chronic illnesses. | 2 years
  With comparable brachial blood pressure ,Do patients with significantly higher central systolic blood pressure have higher risks to have cardiovascular, peripheral arterial and cerebrovascular diseases or not ?

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Univrtsity, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided